CLINICAL TRIAL: NCT06011993
Title: Real-world Analysis on the Efficacy and Safety of Neoadjuvant Therapy for Head and Neck Squamous Cell Carcinoma （neoHNSCC）
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: neoHNSCC
Record Dates: First submitted 2023-08-22; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; Neoadjuvant immunochemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, single-arm study that assesses the efficacy and safety of neoadjuvant immunotherapy combined with platinum-based chemotherapy for Head and Neck Squamous Cell Carcinoma. This trial will also explore the biomarkers of neoadjuvant immunochemotherapy.

DETAILED DESCRIPTION:
This is a retrospective, single-arm study that assesses the efficacy and safety of neoadjuvant immunotherapy combined with platinum-based chemotherapy for Head and Neck Squamous Cell Carcinoma. This trial will also explore the biomarkers of neoadjuvant immunochemotherapy. Patients with untreated, operable, or potentially resectable HNSCC will be included.The pathological results, adverse events and other information of eligible patients will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80, male or female；
* Cytologically or histologically diagnosed squamous cell carcinoma (except mixed squamous cell carcinoma)；
* There was at least one radiographically measurable lesion according to the solid tumor response Evaluation Criteria (RECIST version 1.1)；
* Patients with untreated, operable, or potentially resectable head and neck squamous cell carcinoma；

Exclusion Criteria:

* Malignant diseases other than head and neck squamous cell carcinoma diagnosed within 5 years prior to first administration (excluding basal cell carcinoma of the skin after radical treatment, squamous epithelial carcinoma of the skin, and/or carcinoma in situ after radical resection)；
* Currently participating in an interventional clinical study or has received another investigational drug or has used investigational devices in the 4 weeks prior to initial dosing；
* Evidence of medical history or disease that may interfere with trial results, prevent participants from participating fully in the study, abnormal treatment or laboratory test values, or other conditions that the investigator deems unsuitable for enrollment；

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head and neck squamous cell carcinoma，HNSCC
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 6 months
  Adverse events should be collected, followed up and reported in accordance with prescribed procedures.

SECONDARY OUTCOMES:
Major Pathological Response | 6 months
  MPR, defined as ≤10% of residual surviving tumors
Complete Pathological Response | 6 months
  CPR, defined as no residual survivable tumor cells

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China